CLINICAL TRIAL: NCT05119725
Title: Continuous EKG Monitoring Using S-Patch Ex : Prospective Observational Study (S-patch Registry)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2021-0002
Record Dates: First submitted 2021-10-20; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Patient With Atrial Fibrillation or High Stroke Risk
Keywords: atrial fibrillation; stroke; risk; EKG; continuous
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with atrial fibrillation: Patients with previous diagnosis of atrial fibrillation
  Interventions: Device: continous 3 day EKG monitoring with S-Patch Cardio
- Non-AF patients with high stroke risk: Non-AF patients with high stroke risk
  Interventions: Device: continous 3 day EKG monitoring with S-Patch Cardio

INTERVENTIONS:
Device: continous 3 day EKG monitoring with S-Patch Cardio — continous 3 day EKG monitoring with S-Patch Cardio

SUMMARY:
Atrial fibrillation (AF) is associated with increased mortality and morbidity, and is a dominant, yet preventable, cause of cardioembolic stroke, which has more severe outcomes than other ischaemic stroke causes if left untreated. Approximately 10% of ischemic strokes are associated with AF (AF) first diagnosed at the time of stroke. Detecting asymptomatic AF would provide an opportunity to prevent these strokes by instituting appropriate anticoagulation.

Early diagnosis of AF might enable oral anticoagulant therapy and prevent unwanted consequences of undetected disease, leading to the suggestion that screening for AF might be beneficial in populations at risk. However, there is still debate about whether screen-detected AF bears a similar stroke and mortality risk profile to clinically detected AF, particularly when AF screening is done at a higher intensity than single-time point.

The absence of studies reporting on hard clinical endpoints in AF screening has led to differences in recommendations globally. Most notably, systematic screening for AF is to be considered according to 2020 European guidelines, whereas the US Preventive Services Task Force concluded that current evidence is insufficient to assess the balance of benefits and harms of screening for AF.

The incidence of screen-detected AF strongly depends on the population screened and duration/intensity of screening. Single-time point screening of a general population ≥65 years of age detects undiagnosed AF in 1.4%, and the AF detected is largely persistent. In a large population-based study of individuals 75 to 76 years of age, a more intense 2-week screening program using twice-daily intermittent handheld ECG recordings identified AF in 3.0% (0.5% on the initial ECG4). The identical protocol restricted to those with ≥1 additional stroke risk factor identified 7.4% with AF.

This study was designed in to two arms. The purpose of Arm 1 is to upgrade the artificial intelligence by collecting the continued ECG monitoring data in patients with previous diagnosed AF. The purpose of Arm 2 is to investigate the detection rate of AF using systematic, intensive AF screening with continuous ECG monitoring and the rate of clinical outcome in individuals at high risk during one year follow-up.

DETAILED DESCRIPTION:
Arm 1 Patients with AF are examined with 72 hour continued ECG monitoring Arm 2 Patients with high stroke risk (CHA2DS2-VASc score >=2) are examined with 72 hour continued ECG monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are over the age of 19
2. Those with previous diagnosis of atrial fibrillation
3. Those without atrial fibrillation, but high stroke risk

Exclusion Criteria:

1. Those who refuse to participate in the trial.
2. Those without internet connection

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Referred patients in tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2450 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Number of partipants with atrial fibrillation | At the end of continous ECG monitoring up to 72 hours
  presence of atrial fibrillation

SECONDARY OUTCOMES:
Clinical outcome | 1 year
  composite outcome (all-cause mortality, stroke, transient ischemic accident, systemic embolism, cardiac arrest)
Acquisition rate of ECG | Acquisition rate of ECG signal for 72 hours
  Acquisition rate of ECG signal for 72 hours
Quality of Life | At the enrollment
  Atrial Fibrillation Effect on Quality-of-life (AFEQT) questionnaire: 20 questions, scare from 1 (better outcome) to 7 (worse outcome).
Cognitive function | At the enrollment
  Korean Dementia Screening Questionnaire (KDSQ) questionnaire: 25 questions, scare form 1 (better oucome) to 3 (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SH, Jin JH, Kim J, Lee D, Kim D, Jang J, Yu HT, You SC, Joung B. Wearable device derived electrocardiographic age and its association with atrial fibrillation. NPJ Digit Med. 2026 Jan 17. doi: 10.1038/s41746-026-02344-8. Online ahead of print. PMID 41548032